CLINICAL TRIAL: NCT06772350
Title: Role of Altered Intestinal Permeability and Lipopolysaccharide in Thrombotic Risk and Vascular Injury of Patients With Chronic Inflammatory Bowel Disease
Brief Title: Role of Altered Intestinal Permeability and Lipopolysaccharide in Thrombotic Risk and Vascular Injury in IBD Patients
Acronym: PERVASC-IBD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 7035
Record Dates: First submitted 2024-12-20; First posted 2025-01-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-12

CONDITIONS: IBD
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Experimental
  Interventions: Procedure: examinations

INTERVENTIONS:
Procedure: examinations — Echo-Doppler and blood samples

SUMMARY:
Chronic inflammatory bowel diseases (IBD), including ulcerative colitis (UC) and Crohn's disease (CD), are characterized by chronic immune-mediated inflammation primarily affecting the gastrointestinal tract. Venous and arterial thromboembolic events are significant extra-intestinal manifestations of IBD, but their pathogenic mechanisms are not fully understood. IBD patients have double the risk of venous thromboembolism (VTE) compared to the general population, with particularly high risk in pediatric patients, and an increased mortality rate. They also face a higher risk of early atherosclerosis and future cardiovascular events, such as myocardial infarction, ischemic stroke, and peripheral artery disease. The prevalence of thromboembolic events in IBD ranges from 1.3% to 7.7%, with venous events at around 5% and ischemic heart disease, cerebrovascular disease, and peripheral artery disease at 1-2%.

DETAILED DESCRIPTION:
Chronic inflammatory bowel diseases (IBD), including ulcerative colitis (UC) and Crohn's disease (CD), are characterized by chronic immune-mediated inflammation primarily affecting the gastrointestinal tract. Venous and arterial thromboembolic events are significant extra-intestinal manifestations of IBD, but their pathogenic mechanisms are not fully understood. IBD patients have double the risk of venous thromboembolism (VTE) compared to the general population, with particularly high risk in pediatric patients, and an increased mortality rate. They also face a higher risk of early atherosclerosis and future cardiovascular events, such as myocardial infarction, ischemic stroke, and peripheral artery disease. The prevalence of thromboembolic events in IBD ranges from 1.3% to 7.7%, with venous events at around 5% and ischemic heart disease, cerebrovascular disease, and peripheral artery disease at 1-2%.Several mechanisms contribute to the increased thrombotic risk in IBD, including platelet abnormalities (thrombocytosis and altered platelet function), coagulation factor alterations (e.g., fibrinogen, thrombin), and fibrinolysis defects. Increased oxidative stress and endothelial damage, especially during active disease phases, also play a role. The oxidative stress, caused by reactive oxygen and nitrogen species produced in IBD, leads to molecular and cellular damage, impaired cell homeostasis, and increased mucosal barrier permeability.These changes alone do not fully explain the heightened thrombotic risk in IBD. A reduction in intestinal microbiota diversity and the altered production of metabolites like Trimethylamine-N-oxide (TMAO) may also contribute, along with intestinal permeability changes that allow bacterial products, including lipopolysaccharide (LPS), to enter the bloodstream. LPS, a component of the outer membrane of Gram-negative bacteria, can stimulate low-grade endotoxemia, promoting atherosclerosis and increasing thrombotic risk. Although direct data on this are lacking, these pathological alterations suggest that increased intestinal permeability and circulating LPS may contribute to the elevated venous and arterial thrombotic risk in IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD (both CD and UC, both in active and quiescent stages of disease)
* Age > 18 years
* Signature of informed consent

Exclusion Criteria:

* Other inflammatory states other than IBD (e.g., neoplasm, autoimmune diseases, liver cirrhosis)
* Age < 18 years
* Pregnant woman
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2036-06-15 (Estimated)

PRIMARY OUTCOMES:
Measuring altered intestinal permeability and increased thrombotic risk | 1 year
  altered intestinal permeability will be assessed by measurement of serum LPS and thrombotic risk by echo-Doppler examination

SECONDARY OUTCOMES:
Measuring the relationship between intestinal permeability and how these factors contribute to inflammation and gut microbiota changes in health and disease. | 1 year
  Alteration of intestinal permeability will be assessed by microbiota analysis